CLINICAL TRIAL: NCT02931552
Title: Translating a Stress Management Program for Latinas
Brief Title: Nuevo Amanecer II: Translating a Stress Management Program for Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California Breast Cancer Research Program (Other); National Institute on Aging (NIA) (NIH); Circulo de Vida Cancer Support and Resource Center (Other); Cancer Resource Center of the Desert (Unknown); Family Service Agency of the Central Coast (Unknown); Kaweah Delta Health Care District (Other); San Francisco State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-18737; 21OB-0135 (Other Grant/Funding Number: California Breast Cancer Research Program); 4P30AG015272-20 (NIH)
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Breast Neoplasms; Psychology, Social
Keywords: Breast cancer; Latinas; Peer support counselor; Spanish speaking; Community based; Rural
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nuevo Amancer-II Stress Management Program (Experimental): Nuevo Amanecer-II (NA-II) is a 10-week peer-delivered cognitive-behavioral stress management program. Participants receive the stress management program as soon as possible after randomization.
  Interventions: Behavioral: Nuevo Amancer-II Stress Management Program
- Wait-list Control Group (No Intervention): Waits six months and at the end of the six months is offered the option of receiving the NA-II program.

INTERVENTIONS:
Behavioral: Nuevo Amancer-II Stress Management Program — Participant meets weekly with a trained interventionist called a Compañera (a peer who has had breast cancer) to complete a structured 10-week program designed to develop cognitive and behavioral skills to manage stress and distress, improve communication with family and clinicians, and increase knowledge of self-management after breast cancer.
  Other Names: Nuevo Amanecer II (A New Dawn) cognitive-behavioral stress management program
  Arms: Nuevo Amancer-II Stress Management Program

SUMMARY:
The primary aim is to assess the effectiveness of the Nuevo Amanecer-II (NA-II) cognitive-behavioral stress management program through a 6-month RCT with 150 Spanish-speaking Latinas with breast cancer in three rural settings in terms of improving quality of life (QoL) and reducing distress, compared to a usual care control group (that is offered the program at the end of the 6 months). The investigators will also test the effects of the program on biomarkers of stress (hair and saliva cortisol) and aging (telomere length from saliva). Trained Latinas, called Compañeras (Companions), who have had breast cancer deliver the stress management program in-person to Spanish-speaking Latinas with breast cancer.

DETAILED DESCRIPTION:
The purpose of this study is to adapt Nuevo Amanecer (NA-I) for use in rural populations and test the effects of the new adapted program, NA-II, in a 6-month RCT among 150 rural, low literacy Latinas with non-metastatic breast cancer. Primary outcomes will consist of quality of life and distress. In an ancillary study, the investigators will compare the intervention and wait-list control groups on biomarkers of stress (hair and saliva cortisol) and aging (telomere length from saliva). Finally, to facilitate statewide dissemination of Nuevo Amanecer-II (NA-II), the investigators will develop a guide to implementation for community-based organizations.

The investigators will adapt NA-I to be appropriate for rural and low-literacy Latinas with breast cancer. Needed program adaptations will be identified through a formative evaluation consisting of semi-structured interviews with key informants (e.g., rural Latina breast cancer survivors, advocates, health care providers) and iterative consultations with community representatives in three rural areas with large Latino populations. Results will be applied by the study team and community advisors to adapt NA-I to create NA-II and create the implementation guide.

The investigators will identify key individual, organizational, and community factors that facilitate implementation and support scalability and statewide dissemination through a process evaluation where the investigators will track key implementation activities and debrief program participants, interventionists, and advocates. Products will include NA-II interventionist and participant manuals and a guide to implementation for organizations seeking to replicate the program.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as Latina
* Diagnosed with Stage 0, I, II, or III (non-metastatic) breast cancer
* Primarily Spanish-speaking, or Spanish monolingual
* Aged 18 or older
* Living in surrounding areas of Tulare (Visalia, Dinuba), Santa Cruz (Eastside Santa Cruz, Watsonville, Freedom), or Imperial Valley (El Centro) counties, California.

Exclusion Criteria:

* Terminal illness
* Stage IV breast cancer (distant metastasis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in Physical Well-being Score, a Subscale of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B) | Baseline and 6 month assessment
Change in Social/Family Well-being Score, a Subscale of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B) | Baseline and 6 month assessment
Change Emotional Well-being Score, a Subscale of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B) | Baseline and 6 month assessment
Change in Breast Cancer Concerns Score, a Subscale of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B) | Baseline and 6 month assessment
Change in Functional Well-being Score, a Subscale of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B) | Baseline and 6 month assessment
Change in Total Score of the Functional Assessment of Cancer Therapy-Breast Quality of Life Instrument (FACT-B) | Baseline and 6 month assessment

SECONDARY OUTCOMES:
Change Anxiety Score, a Subscale of the Brief Symptom Inventory (BSI) | Baseline and 6 month assessment
Change Somatization Score, a Subscale of the Brief Symptom Inventory (BSI) | Baseline and 6 month assessment
Change in Personal Health Questionnaire Depression Scale (PHQ-8) Score | Baseline and 6 month assessment
Change Perceived Stress Scale (PSS-10) Score | Baseline and 6 month assessment
Change MOS Health Distress Scale Score | Baseline and 6 month assessment
Change in long-term stress level measured by cortisol levels collected from hair sample. | Baseline and 6 month assessment
  Study staff will collect hair sample pre-intervention (baseline) and at the 6-month follow-up. All hair samples will then be picked up by San Francisco State University Health Equity Research Laboratory (HER) staff for cortisol characterization.
Change in telomere length, a measure of biological aging, in DNA collected from saliva sample. | Baseline and 6 month assessment
  Study staff will collect a saliva sample pre-intervention (baseline) and at the 6-month follow-up. All saliva samples will then be picked up by San Francisco State University Health Equity Research Laboratory (HER) staff to process to extract DNA and measure telomeres.
Change in diurnal cortisol rhythm to assess regulatory patterns through saliva samples collected over 3 days, 3 times/day. | Baseline and 6 month assessment
  Participants will collect nine saliva samples pre-invention (baseline) and at the 6-month follow-up. The first two samples will be taken within the first half hour of waking (first upon awakening and 30 minutes after waking). Participants will collect the last sample right before they go to bed. All saliva samples will then be picked up by San Francisco State University Health Equity Research Laboratory (HER) staff for cortisol characterization.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gregorich, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Multiple Locations, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samayoa C, Santana-Ufret V, Santoyo-Olsson J, Strassle PD, Stewart A, Bonilla J, Escalera C, Mendez RM, Marquez-Magana L, Ortiz C, Ceballos RM, Napoles AM. Cortisol levels in rural Latina breast cancer survivors participating in a peer-delivered cognitive-behavioral stress management intervention: The Nuevo Amanecer-II RCT. Compr Psychoneuroendocrinol. 2022 Jun 24;11:100153. doi: 10.1016/j.cpnec.2022.100153. eCollection 2022 Aug. PMID 35967922
- [Derived] Bonilla J, Alhomsi A, Santoyo-Olsson J, Stewart AL, Ortiz C, Samayoa C, Torres-Nguyen A, Palomino H, Coleman V, Urias A, Gonzalez N, Cervantes SA, Duron Y, Napoles AM. Sharing research results with Latina breast cancer survivors who participated in a community-engaged behavioral RCT study: a descriptive cross-sectional survey study. Trials. 2022 Jan 8;23(1):25. doi: 10.1186/s13063-021-05945-8. PMID 34998436
- [Derived] Bonilla J, Escalera C, Santoyo-Olsson J, Samayoa C, Ortiz C, Stewart AL, Napoles AM. The importance of patient engagement to quality of breast cancer care and health-related quality of life: a cross-sectional study among Latina breast cancer survivors in rural and urban communities. BMC Womens Health. 2021 Feb 9;21(1):59. doi: 10.1186/s12905-021-01200-z. PMID 33563263
- [Derived] Samayoa C, Santoyo-Olsson J, Escalera C, Stewart AL, Ortiz C, Marquez-Magana L, Urias A, Gonzalez N, Cervantes SA, Torres-Nguyen A, Parada-Ampudia L, Napoles AM. Participant-Centered Strategies for Overcoming Barriers to Biospecimen Collection among Spanish-Speaking Latina Breast Cancer Survivors. Cancer Epidemiol Biomarkers Prev. 2020 Mar;29(3):606-615. doi: 10.1158/1055-9965.EPI-19-0942. PMID 32132128